CLINICAL TRIAL: NCT04524000
Title: A Phase II Open-label, 2-Part, Multi-center Study of BYL719 (Alpelisib) in Combination With Fulvestrant for Men and Postmenopausal Women With PIK3CA Mutation Hormone Receptor (HR) Positive, HER2-negative, Advanced Breast Cancer Which Progressed on or After Aromatase Inhibitor (AI) Treatment in Japan
Brief Title: Study Assessing the Efficacy and Safety of Treatment With Alpelisib Plus Fulvestrant in Japanese Men and Postmenopausal Women With Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719C1201
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: HR+; HER2-negative; PIK3CA mutation; Advanced breast cancer; Alpelisib; Fulvestrant; open-label; Part 1; Part 2; Japanese population
MeSH Terms: interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Part 1 of the study has a "Single group" design and the Part 2 has a "Parallel" design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1:CDK4/6 inhibitor naive or pre-treated (Part 1) (Experimental): Participants regardless of prior CDK4/6 inhibitor will be treated at escalating doses (200 mg, 250 mg and 300 mg, orally) of BYL719 in combination with Fulvestrant (500 mg, intramuscular).
  Interventions: Drug: Alpelisib; Drug: Fulvestrant
- Cohort 2: CDK4/6 inhibitor naive (Part 2) (Experimental): Participants who are CDK4/6 inhibitor naive will be treated with BYL719 at the recommended dose identified in Part 1 in combination with Fulvestrant (500 mg, intramuscular).
  Interventions: Drug: Alpelisib; Drug: Fulvestrant
- Cohort 3: CDK4/6 inhibitor pre-treated (Part 2) (Experimental): Participants who are CDK4/6 inhibitor pre-treated will be treated with BYL719 at the recommended dose identified in Part 1 in combination with Fulvestrant (500 mg, intramuscular).
  Interventions: Drug: Alpelisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Alpelisib — [Part 1] Alpelisib administered at 200 mg (DL 1), 250 mg (DL 2) or 300mg (DL 3) orally once daily on a continuous dosing schedule starting on Cycle 1 Day 1 in a 28 day cycle.
  If DL 1 is tolerated, the alpelisib doses of 250 mg will be investigated. If DL 2 is tolerated, the alpelisib doses of 300 mg will be investigated.
  [Part 2] In the Part 2, participants will be enrolled into Cohort 2 (CDK4/6 inhibitor naive) and Cohort 3 (CDK4/6 inhibitor pre-treated) in parallel and alpelisib will be administered at the recommended dose identified in Part 1.
  Other Names: BYL719
Drug: Fulvestrant — Fulvestrant is administered at a dose of 500 mg intramuscular on Cycle 1 Day 1, Day 15, and Day 1 of every cycle thereafter (where a cycle is 28 days).
  Other Names: Faslodex

SUMMARY:
The purpose of this study is to assess the safety and efficacy of alpelisib plus fulvestrant in men and postmenopausal women with hormone receptor (HR) positive, human epidermal growth factor 2 (HER2)-negative, advanced breast cancer harboring a PIK3CA mutation in Japan, whose disease has progressed on or after aromatase inhibitor (AI) treatment regardless of prior CDK4/6 inhibitor use.

DETAILED DESCRIPTION:
This is a Phase II open-label, 2-Part, multi-center study in Japan. The study will be conducted in two parts: Part 1 (Cohort 1) includes participants regardless of prior CDK4/6 inhibitor use and is designed to determine the recommended dose (RD), evaluate the tolerability and safety of alpelisib in combination with fulvestrant. Part 2 consists of 2 cohorts (the CDK4/6 inhibitor naive participants are in Cohort 2 and the CDK4/6 inhibitor pre-treated participants are in Cohort 3) which are designed to assess the efficacy and safety of alpelisib in combination with fulvestrant, will start once the RD of alpelisib is established.

Participants will be treated until disease progression, unacceptable toxicity, death or discontinuation from the study treatment for any other reason and will be followed for survival regardless of treatment discontinuation reason (except if consent is withdrawn or participant is lost to follow up).

ELIGIBILITY:
Inclusion Criteria:

* Japanese man or postmenopausal woman
* Participant has adequate tumor tissue for the analysis of PIK3CA mutational status by a Novartis designated laboratory.
* Participant has identified PIK3CA mutation (as determined by a Novartis designated laboratory)
* Participant has a histologically and/or cytologically confirmed diagnosis of ER+ and/or PgR+ breast cancer by local laboratory
* Participant has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH or SISH) test is required by local laboratory testing
* Participant has measurable disease, i.e., at least one measurable lesion as per RECIST 1.1
* Participant has advanced breast cancer
* Participant has ECOG performance status 0 or 1

Exclusion Criteria:

* Participant with symptomatic visceral disease or any disease burden that makes the participant ineligible for endocrine therapy per the investigator's best judgment
* Participant has received prior treatment;
* with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy), fulvestrant, any PI3K, mTOR or AKT inhibitor for Cohort 1 and 3
* with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy), fulvestrant, any PI3K, mTOR, AKT inhibitor or CDK 4/6 inhibitor for Cohort 2
* Participant has a known hypersensitivity to alpelisib or fulvestrant, or to any of the excipients of alpelisib or fulvestrant
* Participant with inflammatory breast cancer at screening
* Participant is concurrently using other anti-cancer therapy
* Participant has had surgery within 14 days prior to starting study drug or has not recovered from major side effects
* Participant with an established diagnosis at screening of diabetes mellitus type I or not controlled type II (based on FPG and HbA1c)
* Participant has currently documented pneumonitis /interstitial lung disease
* History of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis
* Participant with unresolved osteonecrosis of the jaw
* Participant has a history of severe cutaneous reactions

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
[Part 1] The incidence of Dose Limiting Toxicities (DLTs) of alpelisib in combination with fulvestrant | From Cycle 1 Day 1 to Cycle 2 Day 28 (Cycle = 28 days)
  A DLT is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 2 cycles (the first 56 days) of treatment with alpelisib in combination with fulvestrant and meets any of the criteria specified in the protocol .
[Part 2] Overall Response Rate (ORR) in CDK4/6 inhibitor naive participants | Up to approximately 36 months
  ORR is defined as the proportion of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on local investigator assessment per RECIST 1.1.

SECONDARY OUTCOMES:
[Part 1] Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 37 months
  Safety is determined by incidence, type, and severity of adverse events per CTCAE v4.03 criteria including changes in laboratory values, vital signs, liver assessments, renal and cardiac assessments.
[Part 1] Number of participants with dose adjustments | Up to approximately 37 months
  The number of participants with dose adjustments (reductions, interruption, or permanent discontinuation) and the reasons
[Part 1] Dose intensity for alpelisib and fulvestrant | Up to approximately 37 months
  The dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity)
[Part 1] Duration of exposure for alpelisib and fulvestrant | Up to approximately 37 months
  The duration of exposure (in months) to alpelisib and fulvestrant
[Part 1] Plasma concentrations of alpelisib in combination with fulvestrant | Cycle 1 Day 8 (pre-dose), 15 (pre-dose, post-dose 1 hour, 3 hours) and Day 1 of Cycles 2, 4, 6, 8 (pre-dose) (Cycle = 28 days)
  Summary statistics of alpelisib plasma concentrations by time point and dose level
[Part 2] Overall Response Rate (ORR) for CDK4/6 inhibitor pre-treated participants | Up to approximately 36 months
  ORR is defined as the proportion of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) based on local investigator assessment per RECIST 1.1.
[Part 2] Progression Free Survival (PFS) | Up to approximately 36 months
  PFS is defined as the time from the date of first administration of study treatment until the date of the first documented progression or death due to any cause. PFS will be assessed based on local investigator assessment per RECIST 1.1.
[Part 2] Overall Survival (OS) | Up to approximately 60 months
  OS is defined as the time from date of first administration of study treatment until date of death due to any cause.
[Part 2] Clinical Benefit Rate (CBR) | Up to approximately 36 months
  CBR is defined as the proportion of participants with a best overall response of confirmed CR, or confirmed PR, or an overall response of confirmed stable disease (SD), lasting for a duration of at least 24 weeks. CR, PR, and SD are defined based on local investigator assessment per RECIST 1.1.
[Part 2] Duration of Response (DOR) | Up to approximately 36 months
  DOR only applies to participants whose best overall response is CR or PR based on local investigator assessment per RECIST 1.1. The start date is the date of first documented response of CR or PR (i.e. the start date of response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying cancer.
[Part 2] Time to Response (TTR) | Up to approximately 36 months
  TTR is defined as the time from the date of first administration of study treatment until the date of the first documented response of either CR or PR, which must be subsequently confirmed (although date of initial response is used, not date of confirmation).
[Part 2] Time to definitive deterioration of Eastern Cooperative Oncology Group (ECOG) performance status | Up to approximately 36 months
  Time to definitive deterioration in ECOG performance status is defined as the time from the date of first administration to the date when ECOG performance status has definitively deteriorated by at least one category compared with baseline. Deterioration is considered definitive if there is no subsequent improvement in ECOG performance status back to the baseline category or above.
[Part 2] Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 37 months
  Incidence, type, and severity of adverse events per CTCAE v4.03 criteria including changes in laboratory values, vital signs, liver assessments, renal and cardiac assessments
[Part 2] Number of participants with dose adjustments | Up to approximately 37 months
  The number and percentage of participants with dose interruptions and dose reductions
[Part 2] Dose intensity for alpelisib and fulvestrant | Up to approximately 37 months
  The dose intensity (computed as the ratio of actual cumulative dose received and actual duration of exposure) and the relative dose intensity (computed as the ratio of dose intensity and planned dose intensity)
[Part 2] Duration of exposure for alpelisib and fulvestrant | Up to approximately 37 months
  The duration of exposure (in months) to alpelisib and fulvestrant
[Part 2] Plasma concentrations of alpelisib in combination with fulvestrant | Cycle 1 Day 8 (pre-dose), 15 (pre-dose, post-dose 1 hour, 3 hours) and Day 1 of Cycles 2, 4, 6, 8 (pre-dose) (Cycle= 28 days)
  Summary statistics of alpelisib plasma concentrations by time point and dose level

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Niigata

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com